CLINICAL TRIAL: NCT05913011
Title: Prevalence of Ineffective Esophageal Motility Among Upper Gastrointestinal Symptoms
Brief Title: Prevalence of IEM Among Upper GIT Symptoms
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aya Ahmed Otify, Investigator, Assiut University
Other Study IDs: Prevalence of IEM among U GIT
Record Dates: First submitted 2023-06-12; First posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Esophageal Motility Disorders
MeSH Terms: conditions — Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
* detect the prevalence of IEM among upper git symptom .
* clarify the role of HRM in diagnosis of refractory upper GIT symptoms.

DETAILED DESCRIPTION:
Ineffective esophageal motility (IEM) is characterized by both failed peristalsis and frequent swallows with breaks in the middle/distal peristaltic wave and it may result in symptoms reflecting poor esophageal emptying. As such, IEM may play a role in gastroesophageal reflux disease (GERD) and nonobstructive dysphagia.1 The definition of IEM has evolved after the introduction of high-resolution manometry (HRM), esophageal pressur topography (EPT), and the Chicago Classification of esophageal motility, that-in its second version-defined IEM as weak peristalsis, small (2-5 cm) and large (over 5 cm) peristaltic defects, or frequent (>30%) failed peristalsis. 2 More recently however, the updated third version of the Chicago Classification eliminated small and large breaks from the list of criteria and defined ineffective swallows by a DCI < 45 mmHg.s.cm with ≥50% ineffective swallows constituting IEM, thus eliminating the distinction between failed swallows and weak swallows.3 IEM, as well as fragmented peristalsis, is considered as minor disorders of peristalsis and their clinical significance remains debatable. IEM is the most common abnormality observed in routine esophageal manometry, with an estimated prevalence of 20%-30% reported a prevalence of 51% in patients with esophageal dysphagia. Before 2008 a threshold of 30% was used, but a threshold of 50% correlates better with dysphagia and heartburn.

High-resolution manometry (HRM) provides an improved and more detailed information on esophageal motility when compared to conventional manometry, and today is considered the best test for diagnosis of motility disorders.

ELIGIBILITY:
Inclusion Criteria:

1. patient bove the age of 18 years old
2. All patient presented with upper git symptoms

Exclusion Criteria:

1 - Patients <18 years old 2- patient with known obstructive esophageal disease by endoscopy (i.e. cancer, Stricture) 3- systemic illnesses, scleroderma 4- esophagogastric junction (EGJ) outflow obstruction (mean integrated relaxation pressure ≥15 mmHg).

5- achalasia, 6-Patient who had previouslyundergone esophageal surgery (i.e. antireflux surgery or myotomy) or endoscopic intervention (i.e. transoral fundoplication) were excluded.

7- Patient with atypical (ENT or respiratory) symptoms only . 8-Patient with oropharyngeal dysphagia without associated esophageal symptoms .

9-patient receiving chemotherapy or radiotherapy 10-patient with thyroid disfunction 11- patient with pulber palsy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient bove the age of 18 years old presented with upper git symptoms
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-08 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
detect the prevalence of IEM among upper git symptom | Basline
  detect the prevalence of IEM among upper git symptom
clarify the role of HRM in diagnosis of refractory upper GIT symptoms | Baseline
  clarify the role of HRM in diagnosis of refractory upper GIT symptoms

REFERENCES:
- [Background] Zhuang QJ, Tan ND, Zhang MY, Chen SF, Luo Y, Xiao YL. Ineffective esophageal motility in Chicago Classification version 4.0 better predicts abnormal acid exposure. Esophagus. 2022 Jan;19(1):197-203. doi: 10.1007/s10388-021-00867-5. Epub 2021 Aug 10. PMID 34378104
- [Background] Schlottmann F, Patti MG. Primary Esophageal Motility Disorders: Beyond Achalasia. Int J Mol Sci. 2017 Jun 30;18(7):1399. doi: 10.3390/ijms18071399. PMID 28665309